CLINICAL TRIAL: NCT06537986
Title: Testing the Efficacy of a Neuro-cognitive and Psychosocial Intervention Module in People With Epilepsy
Brief Title: A Neuro-cognitive and Psychosocial Intervention Module in People With Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Neetu Choudhary, Principal Investigator, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12818/PG-20/1 Trg
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Drug Resistant Epilepsy
Keywords: Epilepsy,; Neurocognitive; Psychosocial; module
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Stat Trek software will be adopted to randomize the patients. It is a computer-generated randomization technique. Numbering of the groups has been decided based on coin-flipping.
  1. Intervention group
  2. Control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Standard therapy with intervention module (Module comprised of Cognitive retraining exercise and cognitive behavioral therapy- pen and paper based) Duration - 8 weeks Frequency - once in a week for 2 hours. In person delivery of intervention in a group of 5 patients.
  Interventions: Behavioral: Neurocognitive and psychosocial intervention module
- Control Group (No Intervention): Standard therapy without intervention module

INTERVENTIONS:
Behavioral: Neurocognitive and psychosocial intervention module — The module comprised of various intervention methods that include- I. Cognitive Retraining: Pen-and-paper-based cognitive rehabilitation program that is divided into five hierarchically graded modules: Attention, Visual Processing, Memory, Information Processing, and Executive Functions.
  2.Cognitive-behavioral interventions. Cognitive-behavioral interventions would be carried out for activities scheduling, problem-solving teachings, anger management techniques, modifications of negative cognitions, stigma address measures, and irrational beliefs about epilepsy, etc.
  3. Marital/Family counseling: Marital/family counseling would be done to ensure family understanding of the patient's illness, his/her treatment, prognosis, and outcome. Family complications arising due to illness would also be discussed. Individual and personal needs of the husband, a wife will also be discussed.
  Arms: Intervention Group

SUMMARY:
Patients with epilepsy, especially drug-resistant epilepsy, have a lot of cognitive & psycho-social issues. There is little evidence pertaining to the efficacy of the various cognitive-behavioral interventions and cognitive retraining modules used in epilepsy patients in the Indian context. The real value of these interventions needs further consolidation in terms of its assessment and efficacy. The available literature is scanned and having limitations in terms of assessment tool used, sample size, and also lacks a broader spectrum of psychosocial interventions used. In view of the above limitations, we plan to specially develop & test a Neuro-cognitive and psychosocial intervention module, based on the deficits found in these domains that will help DRE patients to improve their quality of life. This module will be covering not only the broader spectrum of assessment tools but also varieties of interventions. This module will help in planning the future needs of epileptic patients in terms of not only medication but also guide us in choosing the kind of interventions to be used with a particular patient or group of patients.

DETAILED DESCRIPTION:
We plan to specially develop & test a Neuro-cognitive and psychosocial intervention module, based on the deficits found in these domains that will help DRE patients to improve their quality of life. This module will be covering not only the broader spectrum of assessment tools but also varieties of interventions.

AIM To develop and test the efficacy of Neuro-cognitive and psychosocial intervention module in drug-resistant epilepsy.

Clinical Sample: The sample will consist of patients with Drug-resistant epilepsy (DRE). Patients with Drug-resistant epilepsy (DRE) will be included per inclusion and exclusion criteria. The subjects will be taken from the patients attending Refractory epilepsy clinic (REC), Department of Neurology, PGIMER, Chandigarh.

Informed written consent will be obtained from all the study participants per the rules and regulations of the Institutional Ethics Committee of PGIMER.

Study design: It will be a pre and post-design. Subjects fulfilling the inclusion and exclusion criteria will be randomly assigned to intervention and control groups-a Hospital-based Randomized Control Trial Study.

Sample Size: n=60 Follow-up Schedule - Both Pre and post-neuropsychological and psychosocial assessments will be done for all patients.

1. Intervention group - will have an intervention module between pre and post-assessment.
2. Control group - only follow up between Pre and post-assessment. All the randomized patients will be followed up for outcome assessment at 3 to 6 months of the recruitment (Depending on the module).

Statistical Justification:

1. Descriptive statistics will be used in terms of frequency, percentages, range, means, and standard deviations.
2. Group differences between intervention and control groups will be carried out using a t-test.
3. Correlations will be carried out among all the clinical and neuropsychological variables.
4. Linear stepwise regression analysis will be carried out for clinical, neuropsychological, and psychosocial variables separately.
5. Other appropriate statistics would be used as per the requirements of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of 18 - 45 years of age.
2. either gender
3. Willing to participate and sign the informed consent

Exclusion Criteria:

1. Patients with other neurological disorders
2. any other trial at inclusion
3. should not have any major psychiatric disorder
4. pregnant and lactating mothers
5. also, patients who would not be giving informed consent
6. Patients with intellectual disabilities.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2025-01-06 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of improvement in quality of life after receiving an intervention module. | 2 -3 years
  Quality of life in epilepsy-31 scale was used to assess quality of life. The scores are usually transformed into a 0-100 scale, with higher scores indicating a better quality of life.

SECONDARY OUTCOMES:
Evaluation of depression in drug-resistant epilepsy patients after receiving an intervention module. | 2 -3 years
  The Beck Depression Inventory scale was used to assess depression. It is a widely used self-report questionnaire designed to assess the severity of depression in individuals.a total score of 0-13 indicates minimal depression, 14-19 suggests mild depression, 20-28 reflects moderate depression, and a score of 29-63 signifies severe depression.
Evaluation of anxiety in drug-resistant epilepsy patients after receiving an intervention module. | 2 -3 years
  The Hamilton Anxiety Rating Scale was used to assess anxiety. It is a clinician-administered questionnaire used to assess the severity of anxiety symptoms. It consists of 14 items, each rated on a scale from 0 to 4, with higher scores indicating greater anxiety.
Evaluation of stigma in drug-resistant epilepsy patients after receiving an intervention module. | 2 -3 years
  The Stigma Scale of Epilepsy was used to assess stigma. It is a self-report instrument designed to measure perceived stigma among individuals with epilepsy. It is scored by summing the responses to each of its 24 items, which are typically rated on a Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The total score can range from 24 to 96, with higher scores indicating a greater perception of stigma.
Evaluation of Disability in drug-resistant epilepsy patients after receiving an intervention module. | 2 -3 years
  The World Health Organization Disability Assessment Schedule is a standardized instrument for assessing health and disability across various domains. It includes 36 items covering six domains: cognition, mobility, self-care, getting along, life activities, and participation. Each item is rated on a scale from 1 (no difficulty) to 5 (extreme difficulty), and the total score ranges from 36 to 180, with higher scores indicating greater disability.
Evaluation of improvement in attention among patients with drug-resistant epilepsy after receiving an intervention module. | 2 -3 years
  The Trail Making Test (TMT) was used to measure attention. It is a neuropsychological assessment used to measure cognitive flexibility, processing speed, and executive function. It consists of two parts: Part A requires connecting numbered circles in ascending order, while Part B involves alternating between numbers and letters. The time taken to complete each part is recorded, with longer times indicating potential cognitive difficulties. The TMT is commonly used to evaluate cognitive impairments and track changes over time in various clinical and research setting
Evaluation of improvement in memory among patients with drug-resistant epilepsy after receiving an intervention module. | 2 -3 years
  Rey's Auditory Verbal Learning Test was used to assess memory. It is a cognitive assessment designed to evaluate verbal memory and learning abilities. It involves presenting a list of 15 words to the participant, who is asked to recall them immediately after each of five trials. Following these trials, the participant is asked to recall the words after a delay, assessing both short-term and long-term memory. The test also includes a recognition task to evaluate memory accuracy
Evaluation of improvement in executive functioning among patients with drug-resistant epilepsy after receiving an intervention module. | 2 -3 years
  The Wisconsin Card Sorting Test was used to assess executive function. It is a neuropsychological assessment used to evaluate cognitive flexibility, abstract thinking, and executive function. It involves sorting cards based on different categories (color, shape, and number), with the sorting rules changing unpredictably. Participants must adapt to the new sorting rule each time it changes without explicit feedback. Performance is measured by the number of correct responses, errors, and perseverative responses.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Parampreet Singh Kharbanda, MD, DM, Study Chair — PGIMER, Chandigarh
Locations (1):
- Post Graduate institute of medical education and research , Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No